CLINICAL TRIAL: NCT05843656
Title: Enhancing Sleep Dependent Consolidation by Non-invasive Brain Stimulation to Boost Motor Skill Acquisition in Individuals After Stroke
Brief Title: Enhancing Sleep Dependent Consolidation by Non-invasive Brain Stimulation
Acronym: E-ConS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedhelm Hummel (Other)
Responsible Party: Sponsor-Investigator, Friedhelm Hummel, Full Professor, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017-00224
Record Dates: First submitted 2023-03-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Aging
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Slow-wave-like transcranial direct current stimulation (tDCS) (Experimental): tDCS during sleep
  Interventions: Other: Non-invasive brain stimulation
- Spindle-like transcranial alternating current stimulation (tACS) (Experimental): tACS during sleep
  Interventions: Other: Non-invasive brain stimulation
- Sham stimulation during sleep (Sham Comparator): Sham
  Interventions: Other: Non-invasive brain stimulation
- Wake in case participants could not take a nap (Active Comparator): Active Comparator (with stimulation), in case participants could not take a nap
  Interventions: Other: Non-invasive brain stimulation

INTERVENTIONS:
Other: Non-invasive brain stimulation — based on sleep-physiology (slow-wave and spindles)

SUMMARY:
Stroke, one of the most common causes for acquired adult disability, is not only a burden for the individual but also for his or her close relatives and caregivers. Functional recovery is commonly associated with the re-acquisition of lost skills. This skill (re-)acquisition is separated into different phases during which learning takes place while the skill/movement is actively performed - so called online learning - or during the time of non-performance between the training - so called offline learning or consolidation. During the initial phase of training, performance improvements are commonly steep (online learning). During the following processes of consolidation, which often depend on sleep, memory traces are being modified and stored for long-term memory retention leading to a further improvement without additional training (offline learning). Previous studies focusing on individuals after stroke could show a beneficial effect of sleep on motor skill acquisition. As an intervention, transcranial electrical stimulation (tES) with motor tasks could show beneficial effects on motor skill acquisition. tES is a method to stimulate an area of the brain non-invasively and this is done by applying low voltage current to the scalp that lies in close proximity to the target brain region. In the current study, stimulation is performed during sleep and types of stimulation resemble natural sleep physiology: slow-wave and spindles. As slow-wave and spindles are shown to be important for memory consolidation, it is hypothesized that applying physiologically-inspired stimulation could enhance memory consolidation in individuals after stroke. It is known that patterns of sleep physiology change in older individuals, thus, this population is also investigated in the current study. It is interpreted and discussed that older individuals do not benefit from sleep as much as younger individuals do. Thus, it is hypothesized that applying physiologically-inspired stimulation could enhance memory consolidation in healthy older individuals.

ELIGIBILITY:
Inclusion Criteria:

* right handed (healthy older)
* healthy (healthy older)
* monohemispheric stroke (individuals after stroke)
* at least 6 months since diagnosis stroke (individuals after stroke)

Exclusion Criteria:

* Unable to provide informed consent
* Pregnancy
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Non-compliance to the instructions of the experimenter or an inappropriate behaviour hindering the normal progress of the experiment
* Previous enrolment into the current study
* Exclusion criteria tES, and transcranial magnetic stimulation (TMS)
* Use of psychoactive medication, which might influence the study results
* Request of not being informed in case of incidental findings
* Recurrent stroke / multiple strokes (individuals after stroke)
* Cerebellar stroke (individuals after stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-03-19 (Actual)

PRIMARY OUTCOMES:
Behavioural motor score (session 1) | 15 minutes
  It is a computer-based score, which determines (compound) measure of accuracy and speed and can therefore be seen as a measure of performance improvement at session 1
Behavioural motor score (session 2) | 15 minutes
  It is a computer-based score, which determines (compound) measure of accuracy and speed and can therefore be seen as a measure of performance improvement at session 2
Behavioural motor score (session 3) | 15 minutes
  It is a computer-based score, which determines (compound) measure of accuracy and speed and can therefore be seen as a measure of performance improvement at session 3
Behavioural motor score (session 4) | 15 minutes
  It is a computer-based score, which determines (compound) measure of accuracy and speed and can therefore be seen as a measure of performance improvement at session 4

SECONDARY OUTCOMES:
Behavioural motor score (session 5) | 15 minutes
  It is a computer-based score, which determines (compound) measure of accuracy and speed and can therefore be seen as a measure of performance improvement at session 5
Functional magnetic resonance imaging (fMRI) during behavioral motor score evaluation | 15 minutes
  Blood oxygen level dependent contrast among sessions (sessions 1-5)
Electroencephalography (EEG) during sleep | 1 hour
  Sleep spindle density (spindle per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Biotech, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data can be provided/shared upon reasonable request